CLINICAL TRIAL: NCT03258359
Title: A Phase 1 Clinical Trial of Personalized, Adoptive Cellular Immunotherapy Targeting Patient-specific Neoplastic Stem Cell Neoantigens (PACTN) in Patients With Myelodysplastic Syndromes (MDS)
Brief Title: Personalized Adoptive Cellular Therapy Targeting MDS Stem Cell Neoantigens (PACTN)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PersImmune, Inc (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACTN-02
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: MDS
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PACTN (Experimental): Open label 3+3 dose escalation phase 1 trial; 200 to 1000 mL of immunized T cells infused at 0.3, 1, and 3 x 10e7 nucleated cells/kg body weight.
  Interventions: Biological: PACTN

INTERVENTIONS:
Biological: PACTN — To treat patients with MDS who have failed treatment with hypomethylating agents or have relapsed after treatment with hypomethylating agents or have declined hypomethylating therapy.

SUMMARY:
This study will evaluate the safety of autologous T cells that have been immunized ex vivo with patient-specific MDS stem cell neoantigens in patients with MDS.

DETAILED DESCRIPTION:
PACTN is manufactured by a novel method to employ cancer-specific somatic variants (mutations) as a means to immunize autologous T lymphocytes to specifically kill cancer cells bearing the protein products of the mutations.

The PACTN method is based on the premise that somatic DNA mutations that cause cancer often give rise to proteins with an altered amino acid sequence. Peptides derived from these proteins, if expressed in the context of MHC Class I or II may be perceived as "non-self" by the immune system; that is, they may be perceived as neoantigens (aka, neoepitopes). Such neoantigens could therefore serve as immunogenic targets for the development of patient-specific, personalized T cell mediated immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MDS according to the French-American-British (FAB) criteria. Subjects with MDS must have intermediate, high, or very high risk IPSS-R scores and cytopenia of at least one lineage.
* Relapsed/refractory disease, or inadequate response to at least 6 cycles of hypomethylating (HMA) therapy or subjects who decline HMA therapy. Subjects must not have received any MDS or AML directed therapy for >28 days prior to receiving the study treatment.
* Subjects who have opted not to undergo allogeneic hematopoietic stem cell transplantation or for whom no donor is available and who are not deemed eligible for high intensity chemotherapy.
* Age >18 year at the time of obtaining informed consent, male or female.
* An Eastern Cooperative Oncology Grou (ECOG) performance status score of 0, 1, or 2.
* Adequate organ function.
* Seronegative test for HIV-1/2 and hepatitis C antibodies (HCV), and a negative test for Hepatitis B antigen (HBsAg). If hepatitis C antibody test is positive, then the subject must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Women of childbearing potential must have negative pregnancy test prior to initiating study treatment.
* Life expectancy >6 months at time of screening.
* Ability to adhere to the protocol requirements and study visit schedule.

Exclusion Criteria:

* Subjects who anticipate use of other investigational or non-investigational agents for the treatment of MDS during the study period, aside from a stable dose of erythropoietin stimulating agent started >8 weeks prior to screening for this study.
* Subjects who have received investigational agents, cytotoxic chemotherapy, or radiotherapy within 28 days prior to entering the study, or who have not recovered from AEs dur to agents administered more than 28 days earlier.
* Subjects who are less than 21 days from surgery or have insufficient recovery from surgical-related trauma or wound healing.
* Prior history of allogeneic hematopoietic stem cell transplantation.
* Current use of granulocyte colony-stimulating factory (G-CSF) or GM-CSF.
* History of major organ autoimmune disease.
* Concurrent immunosuppressive therapy. A stable dose of prednisone <10 mg daily or inhaled corticosteroids are allowed.
* Any form of primary immunodeficiency.
* Active bacillus tuberculosis (TB) or any other active or uncontrolled infection.
* Pior history of treated malignancy in the past 2 years. Subjects with non-melanoma skin cancer, localized prostate cancer, and carcinoma in situ of the breast of cervix are allowed.
* Impaired cardiac function.
* Pregnant women are excluded from this study as the proposed treatment has not been well studied in pregnant subjects.
* Any other medical or psychiatric disorders, or social situation, that would, in the investigator's opinion, place the subject at unacceptable risk if he/she participates in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute and subacute toxicities and AEs | baseline to four weeks after infusion
  The incidence of dose limiting toxicities (DLTs) after PACTN infusion will be used to determine the maximum tolerated dose (MTD). Adverse effects (AEs) and in particular cytokine release syndrome (CRS) and potential autoimmune AEs will be monitored.

SECONDARY OUTCOMES:
Persistence, abundance, and activity of PACTN | Samples will be collected on days 1, 4, 8, 15, 36, and 57, and then 3, 6, and 12 months
  Determined by quantity of PACTN in the subject's blood sample, assessed by the unique phenotype of PACTN lymphocytes and by functional measurement of PACTN activity (antigen-specific cytotoxicity)
Disease Response | Samples will be collected between day 29 and 43, and then at 3, 6, and 12 months
  Disease response will be assessed by International Working Group (IWG) criteria on bone marrow aspiration
Overall and progression-free survival of subjects who receive PACTN | Six and 12 months after PACTN infusion
  Incidence of subjects who are alive, and both alive and disease - free will be assessed at 6 and 12 months

OTHER OUTCOMES:
The duration of hematologic response, if any | Up to 12 months
  Assessed by measurements of blood counts during subject follow-up, employing IWG criteria
PACTN persistence or peak abundance and clinical response | 6 months and 1 year
  The grouped data on the clinical response and the 6 month and 1-year survival will be analyzed to assess if there is an association between PACTN persistence or peak abundance in blood, and either extent or duration of clinical response or subject survival
Changes in Variant allele frequency (VAF) of somatic mutations targeted by PACTN | From 4 days up to 1 year
  VAFs of targeted mutations will be assessed in blood and marrow after PACTN infusion

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Vitiello, PhD, Study Director — PersImmune, Inc
Locations (1):
- University of California, San Diego, San Diego, California, United States